CLINICAL TRIAL: NCT03629249
Title: A 52-week, Multicenter, Randomized, Double-blind, Double-dummy, Parallel-group, Placebo-controlled Study of Fevipiprant Once Daily Plus Standard-of-care (SoC) for Reduction of Systemic Corticosteroids (Oral and Parenteral) Use in Patients With Severe Asthma
Brief Title: Systemic Corticosteroids Avoidance Study in Severe Asthma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2323; 2018-000212-25 (EudraCT Number)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Obstructive Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity; Immune System Diseases; Fevipiprant; QAW039
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive; Respiratory Hypersensitivity; Hypersensitivity; Immune System Diseases | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QAW039 150 mg (Experimental): QAW039 150 mg once daily orally
  Interventions: Drug: QAW039 150 mg once daily
- QAW039 450 mg (Experimental): QAW039 450 mg once daily orally
  Interventions: Drug: QAW039 450 mg once daily
- Placebo (Placebo Comparator): Placebo to QAW039 once daily orally
  Interventions: Drug: Placebo once daily

INTERVENTIONS:
Drug: Placebo once daily — Placebo to QAW039 once daily (one tablet blinded placebo to QAW039 150 mg and one tablet blinded placebo to QAW039 450 mg).
  Arms: Placebo
Drug: QAW039 150 mg once daily — QAW039 150 mg once daily (one tablet of blinded QAW039 150 mg to be given together with one tablet blinded placebo to QAW039 450 mg)
  Other Names: fevipiprant 150 mg
  Arms: QAW039 150 mg
Drug: QAW039 450 mg once daily — QAW039 450 mg once daily (one tablet of blinded QAW039 450 mg to be given together with one tablet blinded placebo to QAW039 150 mg)
  Other Names: fevipiprant 450 mg
  Arms: QAW039 450 mg

SUMMARY:
The overall purpose of this study was to determine the efficacy of fevipiprant (150 mg and 450 mg once daily), compared with placebo, as add-on to standard-of-care asthma therapy, in terms of avoidance of corticosteroid use over 52 weeks.

DETAILED DESCRIPTION:
This was a randomized, multicenter, double-blind, double-dummy, placebo-controlled, parallel-group study to determine the ability of fevipiprant (QAW039) plus standard-of-care (SoC) compared with placebo plus SoC to reduce the use of systemic corticosteroids (SCS) in patients with severe asthma. The study included:

* a Screening period of up to 2 weeks to assess eligibility;
* a Run-in period of 4 or 10 weeks to evaluate maintenance of asthma control and to collect baseline safety data. The Run-in period was 4 weeks for patients coming with high-dose ICS/LABA (inhaled corticosteroids/long-acting beta-agonist) and 10 weeks for patients switching from mid-dose to high-dose ICS/LABA as per protocol during the run-in period;
* a Treatment period of 52 weeks. Upon completion of the Run-in period, all patients who met eligibility criteria were randomized to 1 of 3 treatment groups (fevipiprant 150 mg or 450 mg or placebo once daily) in a ratio 1:1:1. Randomized patients were stratified according to their peripheral blood eosinophil count (< 250 cells/μl or ≥ 250 cells/μl);
* a Follow-up period of 2 weeks following the last dose of study drug to collect additional data for safety variables.

The main purpose of this study was to determine the efficacy of fevipiprant (150 mg and 450 mg once daily), compared with placebo, as add-on to GINA (Global Initiative for Asthma) treatment step 4 or 5 SoC asthma therapy in terms of avoidance of SCS use over 52 weeks in patients with inadequately controlled severe asthma and high eosinophil counts (eosinophil count at Visit 1 ≥250 cells/ μl) and in the overall patient population regardless of eosinophil counts.

On 16-Dec-2019 the sponsor decided to terminate study CQAW039A2323 earlier than the planned study completion. There were no safety findings with fevipiprant that contributed to this decision. The planned treatment period of 52 weeks was not completed by any patient; patients were treated for a median time of 14 weeks in each group and a maximum of up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of asthma for a period of at least 3 months prior to Screening Visit with current asthma severity step 4 or 5 (GINA 2018)
* Currently on treatment with medium or high dose ICS/LABA +/- other controller (i.e.long-acting muscarinic antagonist (LAMA), leukotriene receptor antagonist (LTRA) etc. as per GINA) for a minimum of 6 weeks prior to Screening Visit
* At screening, patients with FEV1 of ≤80% of the predicted normal value for the patient, after withholding bronchodilators at Screening Visit and beginning of Run-In Visit
* An increase of ≥12% and ≥200 ml in FEV1 approximately 10 to 15 minutes after administration of 400 mcg of salbutamol/albuterol prior to randomization (documented historical reversibility was accepted).
* Demonstration of inadequate control of asthma based on an ACQ-5 score ≥1.5 at Screening Visit and Treatment Day 1 Visit
* Documented history of at least 1 asthma exacerbation within 1 year prior to enrollment

Exclusion Criteria:

* Asthma exacerbation, within 6 weeks prior to enrollment (screening) that required SCS, hospitalization, or emergency room visit
* Chronic/maintenance use of oral corticosteroids (OCS) for asthma (total OCS use days greater than 6 months; continuously or intermittently) within the last year
* Prior use of biologics that has potential to interfere/ affect asthma disease progression, in the previous 6 months from run-in period.
* Any contraindications of SCS use e.g. diabetes, narrow angle glaucoma, or any other as defined by the treating physician
* Pregnant or nursing (lactating) women
* Use of other investigational drugs within 5 half-lives of enrollment, or [within 30 days], whichever is longer

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (96):
- United States (9):
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Westminster, California
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, McKinney, Texas
- Argentina (8):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
- Belgium (4):
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Lebbeke
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Mechelen
- Bulgaria (3):
  - Novartis Investigative Site, Vidin, BGR
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- Chile (2):
  - Novartis Investigative Site, Curicó, Maule Region
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- Colombia (3):
  - Novartis Investigative Site, Zipaquirá, Cundinamarca
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
- Czechia (7):
  - Novartis Investigative Site, Beroun, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Jindřichův Hradec
  - Novartis Investigative Site, Lovosice
  - Novartis Investigative Site, Varnsdorf
- France (4):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Pessac
- Germany (11):
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Witten
- Greece (3):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (10):
  - Novartis Investigative Site, Győr, HUN
  - Novartis Investigative Site, Hajdúnánás, HUN
  - Novartis Investigative Site, Kapuvár, HUN
  - Novartis Investigative Site, Püspökladány, HUN
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Peru (4):
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Cusco
  - Novartis Investigative Site, Lima
  - Novartis Investigative Site, Piura
- Philippines (3):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Iloilo City, Iloilo
  - Novartis Investigative Site, Iloilo City
- Russia (7):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Volgograd
- Slovakia (5):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Spišská Nová Ves, Slovak Republic
  - Novartis Investigative Site, Žilina
- South Africa (2):
  - Novartis Investigative Site, Berea, Durban
  - Novartis Investigative Site, Cape Town
- Spain (4):
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santiago de Compostela
- Novartis Investigative Site, Bangkok, Thailand
- Novartis Investigative Site, Mersin, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, Portsmouth, Hants
  - Novartis Investigative Site, Chertsey, Surrey
  - Novartis Investigative Site, Bradford, West Yorkshire
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 122 investigative sites in 21 countries.
Pre-assignment Details: After the screening, participants went through a Run-in period of 4 or 10 weeks to evaluate maintenance of asthma control and to collect baseline safety data.
Period: Overall Study
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Started (All patients who were randomized) | 201 | 201 | 202
Full Analysis Set (FAS) (All randomized patients who received at least one dose of study medication) | 201 | 200 | 201
Safety Set (SAF) (all patients who received at least one dose of double-blind study drug) | 201 | 200 | 201
Completed | 0 | 0 | 0
Not Completed | 201 | 201 | 202
Not completed — Study terminated by sponsor | 197 | 197 | 194
Not completed — Protocol deviation | 0 | 2 | 5
Not completed — Subject decision | 1 | 1 | 3
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo | Total
Number analyzed (Participants) | 201 | 201 | 202 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.14) | 53.0 (11.99) | 52.8 (12.81) | 53.1 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 136 | 125 | 382
  Male | 80 | 65 | 77 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 180 | 176 | 174 | 530
  Black or African American | 2 | 2 | 2 | 6
  Asian | 10 | 12 | 9 | 31
  American Indian or Alaska Native | 3 | 5 | 13 | 21
  Missing | 6 | 6 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Systemic Corticosteroid Dose in mg Prednisone/Prednisolone or Equivalent Over 52 Weeks in the Overall Population
Description: All participants were provided with prednisone/prednisolone (or equivalent) tablets that could be used according to the asthma plan along with an electronic diary (e-Diary/ePEF). Daily use of oral corticosteroids (number of tablets taken in the previous 12 hours) was recorded once in the morning and once in the evening by the subject in the eDiary/PEF device. In case of use of injectable corticosteroids during certain circumstances (eg. hospitalization) the data was collected on the eCRF (electronic case report form).
  The total systemic corticosteroids (SCS) dose data was aggregated into monthly data for analysis. For the patients discontinuing treatment early, the total SCS dose for 52 weeks was obtained as annualized SCS dose. For example if patient took 120 mg for 3 months then for 12 months patient will be taking 120*12/3=480mg total SCS dose.
  The mean values over 52 weeks in the overall patient population regardless of peripheral blood eosinophil counts are reported here.
Time Frame: 52 weeks
Population: Full Analysis Set (FAS)
Measure: Mean (Full Range); unit: milligrams (mg)
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
milligrams (mg) | 219.67 [0 to 9241.27] | 193.02 [0 to 5184.19] | 223.22 [0 to 9552.69]
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.714, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.734, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Total Systemic Corticosteroid Dose in mg Prednisone/Prednisolone or Equivalent Over 52 Weeks in the Subpopulation of Patients With High Eosinophil Count (≥ 250 Cells/µl)
Description: All participants were provided with prednisone/prednisolone (or equivalent) tablets that could be used according to the asthma plan along with an electronic diary (e-Diary/ePEF). Daily use of oral corticosteroids (number of tablets taken in the previous 12 hours) was recorded once in the morning and once in the evening by the subject in the eDiary/PEF device. In case of use of injectable corticosteroids during certain circumstances (eg. hospitalization) the data was collected on the eCRF (electronic case report form).
  The total systemic corticosteroids (SCS) dose data was aggregated into monthly data for analysis. For the patients discontinuing treatment early, the total SCS dose for 52 weeks was obtained as annualized SCS dose. For example if patient took 120 mg for 3 months then for 12 months patient will be taking 120*12/3=480mg total SCS dose.
  The mean values over 52 weeks in the subpopulation of patients with high peripheral blood eosinophil count at baseline are reported here.
Time Frame: 52 weeks
Population: Participants in the FAS with high peripheral blood eosinophil count count (≥ 250 cells/µl) at baseline
Measure: Mean (Full Range); unit: milligrams (mg)
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 127 | 131 | 127
milligrams (mg) | 210.88 [0 to 5352.80] | 185.29 [0 to 5184.19] | 212.66 [0 to 9552.69]
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.665, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.910, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change From Baseline in Daytime Symptom Scores
Description: All participants were provided with an electronic diary (eDiary/ePEF) to record asthma symptom twice per day. Daytime asthma symptoms were assessed before bed and nighttime asthma symptoms on awakening.
  The daytime asthma symptom score included 4 questions with a range of response categories for each question from 0 to 6 (0 = totally controlled; 6 = extremely poorly controlled). The questions were equally weighted and the overall score (from 0 to 6) was calculated as the average of the 4 questions with higher values indicating more asthma symptoms.
  Mean values of daytime asthma symptom scores were calculated over 4-week intervals during the treatment period.
  The baseline values of daytime asthma symptoms scores were defined as the average score during the run-in period.
  A negative change from baseline in daytime asthma symptom score is a favorable outcome.
Time Frame: Baseline, up to Week 29-32
Population: Participants in the FAS with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
score on scale
  Week 1-4: number analyzed (Participants) | 185 | 184 | 187
  Week 1-4 | -0.12 (0.494) | -0.12 (0.497) | -0.09 (0.459)
  Week 5-8: number analyzed (Participants) | 162 | 155 | 159
  Week 5-8 | -0.21 (0.615) | -0.25 (0.570) | -0.17 (0.561)
  Week 9-12: number analyzed (Participants) | 134 | 133 | 136
  Week 9-12 | -0.29 (0.632) | -0.36 (0.588) | -0.17 (0.605)
  Week 13-16: number analyzed (Participants) | 98 | 96 | 95
  Week 13-16 | -0.32 (0.644) | -0.37 (0.653) | -0.17 (0.629)
  Week 17-20: number analyzed (Participants) | 67 | 68 | 69
  Week 17-20 | -0.30 (0.570) | -0.35 (0.759) | -0.12 (0.622)
  Week 21-24: number analyzed (Participants) | 41 | 34 | 39
  Week 21-24 | -0.31 (0.536) | -0.49 (0.760) | -0.07 (0.688)
  Week 25-28: number analyzed (Participants) | 19 | 17 | 20
  Week 25-28 | -0.13 (0.519) | -0.65 (0.751) | -0.14 (0.726)
  Week 29-32: number analyzed (Participants) | 6 | 4 | 9
  Week 29-32 | -0.54 (0.546) | -0.83 (1.072) | -0.20 (0.887)

4. Secondary Outcome: Change From Baseline in Nighttime Symptom Scores
Description: All participants were provided with an electronic diary (eDiary/ePEF) to record asthma symptom twice per day. Daytime asthma symptoms were assessed before bed and nighttime asthma symptoms on awakening.
  The nighttime asthma symptom score included 1 question with a range of response categories from 0 to 3 (0 = no awakening with asthma symptoms; 3 = awake all night).
  Mean values of nighttime asthma symptom scores were calculated over 4-week intervals during the treatment period.
  The baseline values of nighttime asthma symptoms scores were defined as the average score during the run-in period.
  A negative change from baseline in nighttime asthma symptom score is a favorable outcome.
Time Frame: Baseline, up to Week 29-32
Population: Participants in the FAS with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
score on scale
  Week 1-4: number analyzed (Participants) | 185 | 185 | 188
  Week 1-4 | -0.08 (0.267) | -0.05 (0.281) | -0.07 (0.253)
  Week 5-8: number analyzed (Participants) | 163 | 156 | 159
  Week 5-8 | -0.11 (0.313) | -0.12 (0.314) | -0.13 (0.322)
  Week 9-12: number analyzed (Participants) | 136 | 132 | 135
  Week 9-12 | -0.15 (0.317) | -0.19 (0.369) | -0.12 (0.379)
  Week 13-16: number analyzed (Participants) | 101 | 100 | 96
  Week 13-16 | -0.19 (0.328) | -0.18 (0.360) | -0.12 (0.364)
  Week 17-20: number analyzed (Participants) | 70 | 69 | 69
  Week 17-20 | -0.21 (0.355) | -0.18 (0.397) | -0.17 (0.424)
  Week 21-24: number analyzed (Participants) | 43 | 37 | 41
  Week 21-24 | -0.17 (0.284) | -0.16 (0.323) | -0.14 (0.311)
  Week 25-28: number analyzed (Participants) | 20 | 16 | 20
  Week 25-28 | -0.17 (0.311) | -0.29 (0.355) | -0.15 (0.467)
  Week 29-32: number analyzed (Participants) | 8 | 6 | 9
  Week 29-32 | -0.12 (0.176) | -0.46 (0.505) | -0.24 (0.540)

5. Secondary Outcome: Change From Baseline in ACQ-5 Total Score up to End of Treatment Visit
Description: The Asthma Control Questionnaire (ACQ-5) was completed by the patients at the investigator's site. Patients were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment). The questions were equally weighted and the ACQ-5 score was the mean of the 5 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
  The baseline values of ACQ-5 score were defined as the ACQ-5 scores obtained on Day 1.
  A negative change from baseline in ACQ-5 score is a favorable outcome.
Time Frame: Baseline, up to Week 28
Population: Participants in the FAS with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
score on scale
  Week 6: number analyzed (Participants) | 166 | 158 | 160
  Week 6 | -0.74 (0.852) | -0.94 (0.870) | -0.85 (0.926)
  Week 12: number analyzed (Participants) | 120 | 119 | 119
  Week 12 | -0.97 (0.948) | -1.11 (0.904) | -1.05 (0.884)
  Week 20: number analyzed (Participants) | 60 | 58 | 53
  Week 20 | -1.08 (0.967) | -1.13 (1.075) | -1.22 (0.900)
  Week 28: number analyzed (Participants) | 19 | 13 | 15
  Week 28 | -1.14 (0.943) | -1.52 (1.079) | -1.15 (1.150)

6. Secondary Outcome: Change From Baseline in AQLQ+12 Total Score up to End of Treatment Visit
Description: The Asthma Quality of Life Questionnaire (AQLQ+12) was completed by the patients at the investigator's site. The AQLQ+12 is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to patients with asthma. Patients were asked to recall their experiences during the previous 2 weeks and to score each of the 32 items on a 7-point scale, where 1 indicates maximal impairment and 7 indicates no impairment. Thus, higher scores indicate better asthma-related quality of life. Each item of the AQLQ+12 was equally weighted and the overall score was the mean score of all 32 items and therefore ranged between 1 and 7.
  The baseline values of AQLQ+12 score were defined as the AQLQ+12 scores obtained on Day 1.
  A positive change from baseline in AQLQ+12 score is a favorable outcome.
Time Frame: Baseline, up to Week 28
Population: Participants in the FAS with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
score on scale
  Week 6: number analyzed (Participants) | 166 | 159 | 162
  Week 6 | 0.43 (0.757) | 0.43 (0.762) | 0.40 (0.854)
  Week 12: number analyzed (Participants) | 120 | 119 | 120
  Week 12 | 0.55 (0.884) | 0.60 (0.876) | 0.52 (0.833)
  Week 20: number analyzed (Participants) | 60 | 58 | 53
  Week 20 | 0.64 (0.903) | 0.67 (0.883) | 0.60 (0.867)
  Week 28: number analyzed (Participants) | 19 | 13 | 15
  Week 28 | 0.43 (0.662) | 1.03 (1.178) | 0.55 (1.053)

7. Secondary Outcome: Percentage of Patients Requiring ≥ 7.5 mg Systemic Corticosteroid Dose in mg Prednisone/Prednisolone or Equivalent Per Day Continuously for at Least 30 Days
Description: All participants were provided with prednisone/prednisolone (or equivalent) tablets that could be used according to the asthma plan along with an electronic diary (e-Diary/ePEF) to record medication use. Daily use of oral corticosteroids (the number of tablets taken in the previous 12 hours) was recorded once in the morning and once in the evening by the subject using the eDiary/PEF device. In case of use of injectable corticosteroids during certain circumstances (eg. hospitalization) the data was collected on the eCRF (electronic case report form).
  The percentage of patients requiring ≥ 7.5 mg systemic corticosteroid dose in mg prednisone/prednisolone (or equivalent) per day continuously for at least 30 days within the on-treatment period is presented in this record.
Time Frame: Up to 36 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
Participants | 1 | 0 | 0

8. Secondary Outcome: Percentage of Patients With no Systemic Corticosteroids Use
Description: All participants were provided with prednisone/prednisolone (or equivalent) tablets that could be used according to the asthma plan along with an electronic diary (e-Diary/ePEF) to record medication use. Daily use of oral corticosteroids (the number of tablets taken in the previous 12 hours) was recorded once in the morning and once in the evening by the subject using the eDiary/PEF device. In case of use of injectable corticosteroids during certain circumstances (eg. hospitalization) the data was collected on the eCRF (electronic case report form).
  The percentage of patients with no systemic corticosteroids use up to visit on Week 36 is presented in this record.
Time Frame: Week 36
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
Participants | 170 | 164 | 168

9. Secondary Outcome: Percentage of Patients With Prescription of Biologic Therapy
Description: As part of the flexible therapy, investigators were allowed to prescribe biologics approved for asthma from randomization visit onwards. Prescription of biologic therapy during the treatment period was recorded.
  The proportion of patients with prescription of biologic therapy during the on-treatment period is presented in this record.
Time Frame: Up to 36 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 201 | 200 | 201
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are presented from first dose of study treatment until last dose of study treatment plus 14 days post treatment. Serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, up to maximum duration of 40 weeks.
Description: Any sign or symptom that occurs during the study treatment plus 14 days post treatment for adverse events and 30 days post treatment for serious adverse events.
Groups:
- QAW039 150mg: QAW039 150mg once daily orally
- QAW039 450mg: QAW039 450mg once daily orally
Arm/Group | QAW039 150mg | QAW039 450mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/201 | 0/200 | 0/201
Serious Adverse Events (participants affected / at risk) | 7/201 | 5/200 | 4/201
Other Adverse Events (participants affected / at risk) | 48/201 | 45/200 | 44/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150mg (N=201) | QAW039 450mg (N=200) | Placebo (N=201)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Intentional product misuse (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150mg (N=201) | QAW039 450mg (N=200) | Placebo (N=201)
Nasopharyngitis (Infections and infestations) | 13 | 10 | 13
Asthma (Respiratory, thoracic and mediastinal disorders) | 39 | 41 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT03629249/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03629249/SAP_000.pdf